CLINICAL TRIAL: NCT00965757
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Study of the Combination Therapy of T-614 and Methotrexate in Rheumatoid Arthritis Patients With an Inadequate Response to Methotrexate
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Collaborators: FUJIFILM Toyama Chemical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: T614-ADN
Record Dates: First submitted 2009-08-25; First posted 2009-08-26 (Estimated); Results first posted 2015-06-19 (Estimated); Last update posted 2021-12-17 (Actual); Status verified 2015-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — T 614

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: T-614
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: T-614 — T-614 is administered twice daily in combination with methotrexate. The daily dose of T-614 is 25 mg for the first 4 weeks and 50 mg for subsequent weeks.
  Arms: 1
Drug: Placebo — Placebo is administered twice daily in combination with methotrexate. In placebo group, patients will receive T-614 after completing 28 weeks of treatment.
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of T-614 versus placebo when added to ongoing, stable-dose methotrexate therapy in patients with persistently active rheumatoid arthritis

ELIGIBILITY:
Inclusion criteria:

* Subjects who have a diagnosis of Rheumatoid Arthritis by the ACR criteria
* Age greater or 20 years and less than 70 years old

Exclusion criteria:

* Subject who is considered by the investigator, for any reason, to be an unsuitable candidate for the study
* Women of childbearing potential who are not practicing a successful method of contraception, or wish to become pregnant

Ages: 20 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2009-07-31 (Actual); Primary Completion 2011-09-30 (Actual); Study Completion 2011-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kota Nagai, Study Director — JAC PCU. EPCS, Eisai Co., Ltd.
Locations (72):
- Japan (72):
  - Anjo, Aichi-ken
  - Ichinomiya, Aichi-ken
  - Nagoya, Aichi-ken
  - Okazaki, Aichi-ken
  - Toyohashi, Aichi-ken
  - Ichikawa, Chiba
  - Matsudo, Chiba
  - Narita, Chiba
  - Kitakyushu, Fukuoka
  - Kurume, Fukuoka
  - Maebashi, Gunma
  - Takasaki, Gunma
  - Asahikawa, Hokkaido
  - Chitose, Hokkaido
  - Hakodate, Hokkaido
  - Sapporo, Hokkaido
  - Tomakomai, Hokkaido
  - Amagasaki, Hyōgo
  - Katō, Hyōgo
  - Kobe, Hyōgo
  - Hitachi, Ibaraki
  - Hitachi-Naka, Ibaraki
  - Tsukuba, Ibaraki
  - Kanazawa, Ishikawa-ken
  - Komatsu, Ishikawa-ken
  - Morioka, Iwate
  - Kirishima, Kagoshima-ken
  - Kawasaki, Kanagawa
  - Yokohama, Kanagawa
  - Tamana, Kumamoto
  - Miyagi-gun, Miyagi
  - Sendai, Miyagi
  - Hyūga, Miyazaki
  - Isahaya, Nagasaki
  - Sasebo, Nagasaki
  - Ikoma, Nara
  - Higashiosaka, Osaka
  - Hirakata, Osaka
  - Takatsuki, Osaka
  - Hiki-gun, Saitama
  - Iruma, Saitama
  - Kawaguchi, Saitama
  - Tokorozawa, Saitama
  - Matsue, Shimane
  - Nasushiobara, Tochigi
  - Oyama, Tochigi
  - Shimotsuke, Tochigi
  - Yoshinogawa, Tokushima
  - Chiyoda City, Tokyo
  - Edogawa City, Tokyo
  - Otaku, Tokyo
  - Setagaya City, Tokyo
  - Sumida City, Tokyo
  - Takaoka, Toyama
  - Tonami, Toyama
  - Yonezawa, Yamagata
  - Hōfu, Yamaguchi
  - Fukuoka
  - Gifu
  - Hiroshima
  - Kagashima
  - Kagoshima
  - Kochi
  - Kumamoto
  - Kyoto
  - Nagano
  - Nagasaki
  - Osaka
  - Ōita
  - Saitama
  - Shizuoka
  - Tokushima

RESULTS

PARTICIPANT FLOW:
Groups:
- T-614 (Double-blind, 1-28 Weeks): T-614 was administered in combination with methotrexate. Double blind phase-T-614 was orally administered at dosages of 25 mg/day for the first 4 weeks (25 mg once daily) and 50 mg/day (25 mg twice daily) for subsequent 24 weeks.
- Placebo (Double-blind, 1-28 Weeks): Placebo was administered in combination with methotrexate. Placebo was administered orally at dosages of a tablet once daily for first 4 weeks and a tablet twice daily for subsequent 24 weeks in double-blind period.
- T-614 (Extension, 29-52 Weeks): T-614 was administered in combination with methotrexate. Extension phase- T-614 was orally administered at a dosage of 50 mg/day (25 mg twice daily) for subsequent 24 weeks.
- Placebo/T-614 (Extension, 29-52 Weeks): Participants entered from double-blind placebo phase to 24-week open-label extension phase to receive T-614. T-614 was orally administered at dosages of 25 mg/day for the first 4 weeks (25 mg once daily) and 50 mg/day for subsequent 20 weeks (25 mg twice daily).
Period: Double-blind Phase
Arm/Group | T-614 (Double-blind, 1-28 Weeks) | Placebo (Double-blind, 1-28 Weeks) | T-614 (Extension, 29-52 Weeks) | Placebo/T-614 (Extension, 29-52 Weeks)
Started | 165 | 88 | 0 | 0
Completed | 148 | 70 | 0 | 0
Not Completed | 17 | 18 | 0 | 0
Not completed — Progression of concomitant disease | 1 | 2 | 0 | 0
Not completed — Adverse drug reaction | 2 | 1 | 0 | 0
Not completed — Abnormal Laboratory Value | 2 | 0 | 0 | 0
Not completed — Lack of Efficacy | 7 | 11 | 0 | 0
Not completed — Drug Refusal Due to Adverse Event | 2 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Ineligible after Taking Study Drug | 2 | 3 | 0 | 0
Not completed — Other | 1 | 0 | 0 | 0
Period: Extension Phase
Arm/Group | T-614 (Double-blind, 1-28 Weeks) | Placebo (Double-blind, 1-28 Weeks) | T-614 (Extension, 29-52 Weeks) | Placebo/T-614 (Extension, 29-52 Weeks)
Started | 0 | 0 | 165 | 88
Completed | 0 | 0 | 132 | 64
Not Completed | 0 | 0 | 33 | 24
Not completed — Progression of concomitant disease | 0 | 0 | 4 | 2
Not completed — Adverse drug reaction | 0 | 0 | 6 | 3
Not completed — Abnormal Laboratory Value | 0 | 0 | 6 | 1
Not completed — Lack of Efficacy | 0 | 0 | 8 | 12
Not completed — Drug Refusal Due to Adverse Event | 0 | 0 | 4 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Ineligible after Taking Study Drug | 0 | 0 | 3 | 3
Not completed — Protocol Violation | 0 | 0 | 0 | 1
Not completed — Other | 0 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are presented based on full analysis set, defined as all randomized patients who received at least one dose of study drug and from whom at least one assessment of efficacy under double-blind medication was available.
Groups:
- Total: Total of all reporting groups
Arm/Group | T-614 (Double-blind, 1-28 Weeks) | Placebo (Double-blind, 1-28 Weeks) | Total
Number analyzed (Participants) | 164 | 88 | 252
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.8 (9.9) | 53.5 (10) | 54.3 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 134 | 70 | 204
  Male | 30 | 18 | 48
Duration of Rheumatoid Arthritis [Mean (Standard Deviation); unit: Months] | 53.8 (35) | 50.3 (34) | 52.6 (34.6)

OUTCOME MEASURES:

1. Secondary Outcome: Change From Baseline in Tender Joint Counts and Swollen Joint Counts
Description: Assessment of individual ACR core components like Tender Joint Counts (TJC) and Swollen Joint Counts (SJC)
Time Frame: Week 24 LOCF (for T-614 arm and placebo arm) and Week 52 LOCF (for T614 arm and placebo/T614 arm)
Population: FAS (Double-blind), Efficacy Analysis Set (Extension)
Measure: Mean (Standard Deviation); unit: joint counts
Groups:
- T-614 (Double-blind, 1-28 Weeks) and (Extension, 29-52 Weeks): T-614 was administered in combination with methotrexate. Double blind phase-T-614 was orally administered at dosages of 25 mg/day for the first 4 weeks (25 mg once daily) and 50 mg/day (25 mg twice daily) for subsequent 24 weeks.
  Extension phase- T-614 was orally administered at a dosage of 50 mg/day (25 mg twice daily) for subsequent 24 weeks.
Arm/Group | T-614 (Double-blind, 1-28 Weeks) and (Extension, 29-52 Weeks) | Placebo (Double-blind, 1-28 Weeks) | Placebo/T-614 (Extension, 29-52 Weeks)
Number analyzed (Participants) | 164 | 88 | 68
joint counts
  Baseline: TJC | 12.5 (6.5) | 13.3 (8.1) | 13.8 (8.5)
  Change from baseline at week 24 LOCF: TJC | -7.4 (6) | -4.6 (7.8) | NA (NA) — Week 24 is not applicable as this arm starts from week 29 to week 52
  Change from baseline at week 52 LOCF: TJC | -8.4 (6.1) | NA (NA) — Week 52 is not applicable as this arm completed at week 28 | -9.9 (7.6)
  Baseline: SJC | 11.5 (6.3) | 11.1 (5.7) | 10.9 (5.8)
  Change from baseline at week 24 LOCF: SJC | -6.5 (5.9) | -2.9 (6.7) | NA (NA) — Week 24 is not applicable as this arm starts from week 29 to week 52
  Change from baseline at week 52 LOCF: SJC | -7.1 (6.8) | NA (NA) — Week 52 is not applicable as this arm completed at week 28 | -6.3 (6.5)

2. Secondary Outcome: Change From Baseline in PAP, PtGADA and PyGADA
Description: Patient's assessment of pain (PAP), patient's global assessment of disease activity (PtGADA) and physician's global assessment of disease activity (PyGADA) each was assessed on a visual analog scale ranging from 0-100 mm, with higher scores indicating severe disease.
Time Frame: Week 24 LOCF (for T-614 arm and placebo arm) and Week 52 LOCF (for T614 arm and placebo/T614 arm)
Population: FAS (Double-blind), Efficacy Analysis Set (Extension)
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | T-614 (Double-blind, 1-28 Weeks) and (Extension, 29-52 Weeks) | Placebo (Double-blind, 1-28 Weeks) | Placebo/T-614 (Extension, 29-52 Weeks)
Number analyzed (Participants) | 164 | 88 | 68
mm
  Baseline PAP | 47.5 (22.2) | 46.4 (23.1) | 44.8 (22.4)
  Change from baseline in PAP: week 24 LOCF | -22 (23.8) | -2.5 (27) | NA (NA) — Week 24 is not applicable as this arm starts from week 29 to week 52
  Change from baseline in PAP: week 52 LOCF | -24 (24.1) | NA (NA) — Week 52 is not applicable as this arm completed at week 28 | -21.4 (26.6)
  Baseline PtGADA | 47.7 (24.3) | 50.1 (23.5) | 48.4 (23.6)
  Change from baseline in PtGADA: week 24 LOCF | -21.2 (26.4) | -5 (27.1) | NA (NA) — Week 24 is not applicable as this arm starts from week 29 to week 52
  Change from baseline in PtGADA: week 52 LOCF | -24.3 (26) | NA (NA) — Week 52 is not applicable as this arm completed at week 28 | -23.1 (27.7)
  Baseline PyGADA | 52.6 (18.3) | 53.2 (19) | 52.1 (17.9)
  Change from baseline in PyGADA: week 24 LOCF | -27.1 (19.3) | -10.4 (26.6) | NA (NA) — Week 24 is not applicable as this arm starts from week 29 to week 52
  Change from baseline in PyGADA: week 52 LOCF | -29.1 (22.4) | NA (NA) — Week 52 is not applicable as this arm completed at week 28 | -29.9 (24.4)

3. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire Disability Index (HAQ-DI)
Description: HAQ-DI was a participant assessed measure of health assessment, measured on a single scale ranging from 0 (no difficulty) to 3 (unable to do), with higher scores indicating severe disease.
Time Frame: Week 24 LOCF (for T-614 arm and placebo arm) and Week 52 LOCF (for T614 arm and placebo/T614 arm)
Population: FAS (Double-blind), Efficacy Analysis Set (Extension)
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | T-614 (Double-blind, 1-28 Weeks) and (Extension, 29-52 Weeks) | Placebo (Double-blind, 1-28 Weeks) | Placebo/T-614 (Extension, 29-52 Weeks)
Number analyzed (Participants) | 164 | 88 | 68
score on scale
  Baseline | 0.8178 (0.5525) | 0.7344 (0.5117) | 0.7188 (0.5274)
  Week 24 LOCF | -0.3544 (0.4492) | 0.0256 (0.549) | NA (NA) — Week 24 is not applicable as this arm starts from week 29 to week 52
  Week 52 LOCF | -0.4093 (0.4566) | NA (NA) — Week 52 is not applicable as this arm completed at week 28 | -0.2904 (0.4669)

4. Secondary Outcome: Change From Baseline in C-reactive Protein (CRP)
Description: Assessment of individual ACR core components i.e. CRP
Time Frame: Week 24 LOCF (for T-614 arm and placebo arm) and Week 52 LOCF (for T614 arm and placebo/T614 arm)
Population: FAS (Double-blind), Efficacy Analysis Set (Extension)
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | T-614 (Double-blind, 1-28 Weeks) and (Extension, 29-52 Weeks) | Placebo (Double-blind, 1-28 Weeks) | Placebo/T-614 (Extension, 29-52 Weeks)
Number analyzed (Participants) | 164 | 88 | 68
mg/dl
  Baseline | 1.843 (1.943) | 1.705 (1.583) | 1.714 (1.611)
  Week 24 LOCF | -0.528 (2.067) | 0.47 (2.028) | NA (NA) — Week 24 is not applicable as this arm starts from week 29 to week 52
  Week 52 LOCF | -0.609 (1.841) | NA (NA) — Week 52 is not applicable as this arm completed at week 28 | -0.581 (1.866)

5. Secondary Outcome: Change From Baseline in Erythrocyte Sedimentation Rate (ESR)
Description: Assessment of individual ACR core components i.e. ESR
Time Frame: Week 24 LOCF (for T-614 arm and placebo arm) and Week 52 LOCF (for T614 arm and placebo/T614 arm)
Population: FAS (Double-blind), Efficacy Analysis Set (Extension)
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | T-614 (Double-blind, 1-28 Weeks) and (Extension, 29-52 Weeks) | Placebo (Double-blind, 1-28 Weeks) | Placebo/T-614 (Extension, 29-52 Weeks)
Number analyzed (Participants) | 164 | 88 | 68
mm/hr
  Baseline | 45.6 (21) | 41.8 (22.5) | 40.1 (23.2)
  Week 24 LOCF | -9.3 (20.8) | 2.6 (19.7) | NA (NA) — Week 24 is not applicable as this arm starts from week 29 to week 52
  Week 52 LOCF | -9.4 (21.3) | NA (NA) — Week 52 is not applicable as this arm completed at week 28 | -8.8 (21.5)

6. Secondary Outcome: Disease Activity Score in 28 Joints (DAS28): The Rates of Remission (DAS28-CRP Less Than 2.6), and Low Disease Activity (DAS28-CRP Less Than 3.2)
Description: The DAS28 is a composite score derived from 4 of these measures i.e count of 28 swollen joints, 28 tender joints, measure erythrocyte sedimentation rate (ESR) or C reactive protein (CRP) and to make a 'global assessment of health' (indicated by marking a 10 cm line between very good and very bad). DAS28 is assessed as score on scale from 0 to 10 indicating current rheumatoid arthritis (RA) disease activity (0= low disease activity and 10 = high disease activity).
Time Frame: Week 24 LOCF (for T-614 arm and placebo arm) and Week 52 LOCF (for T614 arm and placebo/T614 arm)
Population: FAS (Double-blind), Efficacy Analysis Set (Extension)
Measure: Number; unit: participants
Arm/Group | T-614 (Double-blind, 1-28 Weeks) and (Extension, 29-52 Weeks) | Placebo (Double-blind, 1-28 Weeks) | Placebo/T-614 (Extension, 29-52 Weeks)
Number analyzed (Participants) | 164 | 88 | 68
participants
  Remission: week 24 LOCF | 45 | 8 | NA — Week 24 is not applicable as this arm starts from week 29 to week 52
  Remission: week 52 LOCF | 56 | NA — Week 52 is not applicable as this arm completed at week 28 | 23
  Low Disease Activity: week 24 LOCF | 78 | 18 | NA — Week 24 is not applicable as this arm starts from week 29 to week 52
  Low Disease Activity: week 52 LOCF | 88 | NA — Week 52 is not applicable as this arm completed at week 28 | 38

7. Secondary Outcome: Percentage of ACR 50 Criteria Responders
Description: ACR50 response is defined as at least a 50% improvement in tender joint count and swollen joint count, and in three of five of the following measures: patient pain intensity assessment, patient global assessment, physician global assessment, Health assessment questionnaire disability index (HAQ-DI), and an acute phase reactant [erythrocyte sedimentation rate (ESR) or C-reactive protein (CRP)].
Time Frame: Week 24 LOCF (for T-614 arm and placebo arm) and Week 52 LOCF (for T614 arm and placebo/T614 arm)
Population: Full Analysis Set (Double-blind), Efficacy Analysis Set (Extension)
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | T-614 (Double-blind, 1-28 Weeks) and (Extension, 29-52 Weeks) | Placebo (Double-blind, 1-28 Weeks) | Placebo/T-614 (Extension, 29-52 Weeks)
Number analyzed (Participants) | 164 | 88 | 68
Percentage of Participants
  Week 24 LOCF | 38.4 [30.9 to 46.3] | 15.9 [9 to 25.2] | NA [NA to NA] — Week 24 is not applicable as this arm starts from week 29 to week 52
  Week 52 LOCF | 49.4 [41.5 to 57.3] | NA [NA to NA] — Week 52 is not applicable as this arm completed at week 28 | 45.6 [33.5 to 58.1]

8. Secondary Outcome: Percentage of ACR 70 Criteria Responders
Description: ACR70 response is defined as at least a 70% improvement in tender joint count and swollen joint count, and in three of five of the following measures: patient pain intensity assessment, patient global assessment, physician global assessment, Health assessment questionnaire disability index (HAQ-DI), and an acute phase reactant [erythrocyte sedimentation rate (ESR) or C-reactive protein (CRP)].
Time Frame: Week 24 LOCF (for T-614 arm and placebo arm) and Week 52 LOCF (for T614 arm and placebo/T614 arm)
Population: FAS (Double-blind), Efficacy Analysis Set (Extension)
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | T-614 (Double-blind, 1-28 Weeks) and (Extension, 29-52 Weeks) | Placebo (Double-blind, 1-28 Weeks) | Placebo/T-614 (Extension, 29-52 Weeks)
Number analyzed (Participants) | 164 | 88 | 68
Percentage of Participants
  Week 24 LOCF | 17.1 [11.7 to 23.7] | 5.7 [1.9 to 12.8] | NA [NA to NA] — Week 24 is not applicable as this arm starts from week 29 to week 52
  Week 52 LOCF | 23.8 [17.5 to 31] | NA [NA to NA] — Week 52 is not applicable as this arm completed at week 28 | 22.1 [12.9 to 33.8]

9. Primary Outcome: Percentage of American College of Rheumatology [ACR] 20 Criteria Responders
Description: ACR20 response is defined as at least a 20% improvement in tender joint count and swollen joint count, and in three of five of the following measures: patient pain intensity assessment, patient global assessment, physician global assessment, Health assessment questionnaire disability index (HAQ-DI), and an acute phase reactant [erythrocyte sedimentation rate (ESR) or C-reactive protein (CRP)].
Time Frame: Week 24 Last Observation Carried Forward (LOCF) (for T-614 arm and placebo arm) and Week 52 LOCF (for T-614 arm and placebo/T614 arm)
Population: Full Analysis Set (Double-blind), Efficacy Analysis Set (Extension)
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | T-614 (Double-blind, 1-28 Weeks) and (Extension, 29-52 Weeks) | Placebo (Double-blind, 1-28 Weeks) | Placebo/T-614 (Extension, 29-52 Weeks)
Number analyzed (Participants) | 164 | 88 | 68
Percentage of Participants
  Week 24 LOCF | 69.5 [61.9 to 76.5] | 30.7 [21.3 to 41.4] | NA [NA to NA] — Week 24 is not applicable as this arm starts from week 29 to week 52
  Week 52 LOCF | 71.3 [63.8 to 78.1] | NA [NA to NA] — Week 52 is not applicable as this arm completed at week 28 | 72.1 [59.9 to 82.3]

ADVERSE EVENTS:
Time Frame: Up to 1 - 52 weeks for T614 (double-blind and extension) arm, up to 1 - 24 weeks for placebo (double-blind) arm and Up to 29 - 52 Weeks for placebo/T614 (extension) arm.
Description: Treatment emergent adverse events are presented in this section.
Arm/Group | T-614 (Double-blind, 1-28 Weeks) and (Extension, 29-52 Weeks) | Placebo (Double-blind, 1-28 Weeks) | Placebo/T-614 (Extension, 29-52 Weeks)
Serious Adverse Events (participants affected / at risk) | 2/164 | 2/88 | 0/68
Other Adverse Events (participants affected / at risk) | 135/164 | 43/88 | 41/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | T-614 (Double-blind, 1-28 Weeks) and (Extension, 29-52 Weeks) (N=164) | Placebo (Double-blind, 1-28 Weeks) (N=88) | Placebo/T-614 (Extension, 29-52 Weeks) (N=68)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Gastroduodenal ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Fallopian tube cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cardiac Failure (Cardiac disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | T-614 (Double-blind, 1-28 Weeks) and (Extension, 29-52 Weeks) (N=164) | Placebo (Double-blind, 1-28 Weeks) (N=88) | Placebo/T-614 (Extension, 29-52 Weeks) (N=68)
Nasopharyngitis (Infections and infestations) | 52 (71) | 14 (18) | 15 (17)
Pharyngitis (Infections and infestations) | 10 (14) | 6 (6) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 20 (25) | 2 (3) | 4 (4)
Stomatitis (Gastrointestinal disorders) | 18 (26) | 2 (2) | 4 (4)
Lymphocyte count decreased (Investigations) | 29 (48) | 8 (13) | 7 (12)
Aspartate aminotransferase increased (Investigations) | 27 (44) | 5 (5) | 3 (4)
Alanine aminotransferase increased (Investigations) | 24 (31) | 7 (7) | 5 (6)
Beta 2 microglobulin increased (Investigations) | 15 (17) | 2 (2) | 5 (5)
Beta 2 microglobulin urine increased (Investigations) | 15 (20) | 1 (1) | 4 (7)
Blood iron decreased (Investigations) | 43 (71) | 16 (26) | 9 (10)
Bronchitis (Infections and infestations) | 8 (10) | 0 (0) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 11 (13) | 0 (0) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 8 (9) | 0 (0) | 4 (5)
Rash (Skin and subcutaneous tissue disorders) | 9 (10) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (11) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 15 (19) | 0 (0) | 2 (3)
Blood urea increased (Investigations) | 13 (16) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other